CLINICAL TRIAL: NCT00013702
Title: Adefovir Dipivoxil for the Treatment of Hepatitis B in Human Immunodeficiency Virus Infected Patients With Decompensated Hepatitis B Liver Disease and a Hepatitis B Viral Load of at Least 1.0 X 10(6) (Copies/mL) Despite 52 Weeks of Lamivudine Therapy
Brief Title: Adefovir Dipivoxil to Treat Hepatitis B in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010134; 01-I-0134
Record Dates: First submitted 2001-03-28; First posted 2001-03-29 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-02

CONDITIONS: Hepatitis B; HIV Infection
Keywords: Immunology; Cirrhosis; Ascites; Open-Label; Chronic; HIV; Hepatitis B
MeSH Terms: conditions — Hepatitis B; HIV Infections; Fibrosis; Ascites; Bronchiolitis Obliterans Syndrome | interventions — adefovir

INTERVENTIONS:
Drug: Adefovir

SUMMARY:
This study will evaluate the safety and effectiveness of adding the experimental drug adefovir dipivoxil to lamivudine for treating hepatitis B virus (HBV) infection in HIV-infected patients with liver cirrhosis. Adefovir inhibits HBV by interfering with replication of the virus's genetic material. In some people, the drug has been active against strains of HBV that are resistant to lamivudine; it may also have some activity against HIV.

HIV-infected patients 21 years of age and older with chronic hepatitis B infection and liver cirrhosis who have received lamivudine treatment for at least 1 year may be eligible for this 48-week study. Candidates will be screened with a complete medical history, blood tests and a 24-hour urine collection. Blood tests include HLA typing (a test of genetic markers on white blood cells that permit specialized immunology studies). Within 4 weeks, candidates who appear eligible for the study will have a physical examination and medical history, an abdominal ultrasound (imaging test using sound waves) to check for cancer of the liver, chest X-ray and electrocardiogram (EKG). Blood and urine tests will also be done, and women who can become pregnant will have a pregnancy test.

Patients who meet the study criteria and decide to participate will then start treatment with one 10-mg adefovir pill per day by mouth. In addition, patients will continue to take all other medications prescribed by their doctor. Follow-up clinic visits will be scheduled as follows:

* Days 1, 3, 5, 7, 10 and 21 - Blood will be drawn for specialized immunology tests and to measure blood levels of HIV and HBV.
* Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 - Blood and urine (single sample) tests will be done to determine the side effects of adefovir and its effect on the HBV infection.
* Week 48 or early termination (end of study) - Blood tests (including tests for hepatitis C and D), abdominal ultrasound and a 24-hour urine collection to evaluate kidney function will be done.
* Monthly visits beyond week 48 - Based on the HBV response to treatment and the availability of the drug from the sponsor, patients may be offered to extend their treatment with adefovir. Those who continue will have monthly follow-up visits for blood and urine (single sample) tests.

DETAILED DESCRIPTION:
Patients co-infected with human immunodeficiency virus (HIV) and hepatitis B virus (HBV) who have advanced liver disease (decompensated cirrhosis by Child-Pugh score and no known cause of hepatitis other than HBV), a HBV viral load of at least 1 million copies/mL blood, and at least one year of therapy with lamivudine will be treated with open-label adefovir dipivoxil 10 mg daily and lamivudine 150 mg bid to evaluate the safety and efficacy of this regimen in this patient group and to obtain specimens for studies of immune responses to HBV in HIV-infected patients. Additionally the kinetics of viral load response to adefovir will be assessed. Specimens will be stored for possible use in evaluating HBV and HIV resistance to adefovir. L-carnitine supplementation will be used only if low serum carnitine levels are documented. Patients will be followed for HBV viral load response to adefovir for 48 weeks with possible extension. The primary study endpoints will be HBV viral load at week 24 (per-protocol patients) and DAVG at week 24 (intent-to-treat patients). Adefovir will be discontinued for toxicity; there will be no dose reduction. Up to 30 subjects will be enrolled.

ELIGIBILITY:
INCLUSION CRITERIA:

Age greater than or equal to 18 years

Infection with HBV with HBV viral load greater than or equal to 1.0 x 10(6) copies/mL by Roche assay at screen

HIV-infected as documented by ELISA and Western Blot in NIAID clinic (any CD4/HIV viral load)

Decompensated cirrhosis (Child-Pugh Score greater than or equal to 7: Class B or C cirrhosis)

Class A with Score of 6 acceptable if secondary to ascites grading and not encephalopathy or laboratory abnormality (PT, albumin, bilirubin).

Able to return to NIH for study visits

Have a physician(s) outside of NIH who will provide routine, as well as HIV and liver specific, care.

Receiving lamivudine at a dose of at least 100 mg qd for greater than or equal to one year prior to enrollment (with no dosing interruptions of greater than 1 month total in the previous year and no interruption in the 3 months prior to study entry)

Serum creatinine less than 1.5 mg/dL

Serum phosphorus greater than or equal to 2.2 mg/dL (normal range NIH 2.3-4.3 mg/dL)

Neutrophil count greater than or equal to 1000 cells/mm(3)

Platelets greater than or equal to 50,000/mm(3)

Hemoglobin greater than or equal to 8.0 mg/dL

ALT less than or equal to 287 (7 X the NIH upper limit of normal)

Not pregnant or breast-feeding. Pregnancy test must be negative within two weeks prior to dosing with study medications.

If capable of pregnancy: use of effective contraception during study: effective contraception methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap or sponge, or use of hormonal contraception with an anti-HIV regimen that will not alter metabolism of hormonal contraception

Willing and able to provide written informed consent

Because liver disease can result in encephalopathy, willing to designate a person for durable power of attorney on the NIH form for medical research and medical care purposes at the NIH Clinical Center

EXCLUSION CRITERIA:

Prior use of ADV (outside of patient receiving adefovir from NIH under emergency use IND) or prior use of tenofovir, or cidofovir

Active serious systemic infections other than HIV or HBV

Liver disease caused by reasons other than hepatitis B e.g., HCV, HDV, Wilson's, hemochromatosis, autoimmune hepatitis (ANA greater than or equal to 160) except history of drug-associated hepatitis with discontinuation of causative agent

History of significant encephalopathy

History of clinically significant pancreatitis

History of untreated varices

New AIDS-defining event other than esophageal candidiasis diagnosed within one month prior to baseline

Decompensated heart failure

Treatment with immunomodulator drugs (interferons, interleukins, corticosteroids in greater than physiologic doses) in the 4 weeks prior to baseline. G-CSF and epoietin use are permitted.

Anti-HBV therapy other than lamivudine (such as emtricitabine, lobucavir, entecavir, HBIG, clevudine, MCC-478) with the exception of interferon alpha, famciclovir or foscarnet that ended more than 12 weeks prior to screen.

Hepatic mass suggestive of hepatocellular carcinoma

Alpha-fetoprotein level greater than or equal to 200ng/mL

Evidence of gastrointestinal malabsorption or chronic nausea or vomiting

Current alcohol or substance abuse that potentially could interfere with patient compliance

Malignancy other than cutaneous Kaposi's sarcoma, skin cancer treated by resection or HPV-associated carcinoma in situ or Bowen's disease in the 5 years prior to enrollment

History of clinically significant renal dysfunction within the previous 12 months prior to baseline

Concomitant therapy with aminoglycosides, amphotericin B, cidofivir, cisplatinum, IV pentamidine, vancomycin, systemic chemotherapeutic agents, probenecid or other nephrotoxic agents

Proteinuria (greater than or equal to 3+)

ANA greater than or equal to 3 EU

Positive PCR test for hepatitis C

Antibodies to hepatitis D (delta hepatitis)

Pregnancy or breast-feeding

History of organ or bone marrow transplantation

Any systemic illness that will make it unlikely that the subject will be able to return to NIH for the required study visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2001-03; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Colin JF, Cazals-Hatem D, Loriot MA, Martinot-Peignoux M, Pham BN, Auperin A, Degott C, Benhamou JP, Erlinger S, Valla D, Marcellin P. Influence of human immunodeficiency virus infection on chronic hepatitis B in homosexual men. Hepatology. 1999 Apr;29(4):1306-10. doi: 10.1002/hep.510290447. PMID 10094979
- [Background] Honkoop P, de Man RA, Niesters HG, Zondervan PE, Schalm SW. Acute exacerbation of chronic hepatitis B virus infection after withdrawal of lamivudine therapy. Hepatology. 2000 Sep;32(3):635-9. doi: 10.1053/jhep.2000.16333. PMID 10960461
- [Background] Lai CL, Chien RN, Leung NW, Chang TT, Guan R, Tai DI, Ng KY, Wu PC, Dent JC, Barber J, Stephenson SL, Gray DF. A one-year trial of lamivudine for chronic hepatitis B. Asia Hepatitis Lamivudine Study Group. N Engl J Med. 1998 Jul 9;339(2):61-8. doi: 10.1056/NEJM199807093390201. PMID 9654535